CLINICAL TRIAL: NCT04431024
Title: Prospective Evaluation of High Resolution Dual Energy Computed Tomographic Imaging, Noninvasive (Liquid) Biopsies, and Minimally Invasive Surgical Surveillance for Early Detection of Mesotheliomas in Patients With BAP1 Tumor Predisposition Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200106; 20-C-0106
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12-16

CONDITIONS: Familial Cancer; BRCA1-Associated Protein-1 (BAP1) Mutations; Tumor Predisposition Syndrome (TPDS); Mesothelioma
Keywords: Germline Mutation in the BAP1 Gene; BRCA1-Associated Protein-1; Genetics; Familial Background; Natural History; DECT
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients: Individuals with history of cancer and detected or suspected germline mutation in BAP1 TPDS
- Relatives of cancer patients: First- or second-degree relatives of a cancer patient (with or without cancer) with documented BAP1 tumor predisposition syndrome (TPDS)

SUMMARY:
Background:

A germline mutation is a change to a person s genes that is carried through their DNA. These mutations can be passed on from parents to their offspring. Germline mutations in a gene called BAP1 are linked to the development of mesothelioma and other cancers. Researchers want to follow people with these mutations to learn more.

Objective:

To see if researchers can improve how people who have or are suspected to have a BAP1 mutation are monitored over time.

Eligibility:

People age 30 and older who are suspected to have a BAP1 germline mutation.

Design:

Participants will be screened with a personal and family medical history. Their medical records may be reviewed. They will give a blood or saliva sample to test for a BAP1 mutation. They will get genetic counseling.

To take part in this study, participants will enroll on 2 to 3 other protocols.

Participants will have a physical exam. They may have a tumor biopsy. They will give blood and urine samples. They will have skin and eye exams.

Some participants will have video-assisted thoracoscopy to examine the chest and lungs and diagnose suspicious areas. For this, a small camera is inserted into the chest through a small incision.

Some participants will have laparoscopy to examine the organs inside the abdomen. For this, a small camera is inserted into the abdomen through a small incision.

Participants will have imaging scans of the chest, abdomen, and pelvis. They may have brain scans.

Participants will visit the NIH once a year for follow-up exams.

Participation lasts indefinitely.

DETAILED DESCRIPTION:
Background:

* Mutations involving BRCA1-Associated Protein-1 (BAP1), a nuclear deubiquitinase involved in epigenetic regulation of gene expression, DNA repair, and cellular energetics, have emerged as one of the most common somatic mutations in malignant mesotheliomas.
* Germline mutations involving BAP1 predispose individuals to mesothelioma as well as a variety of other malignancies including melanoma and lung, renal, gastric, breast, and biliary tract cancers.
* The cancer penetrance of germline BAP1 mutations is nearly 100%, with most patients developing multiple neoplasms.
* Presently there are no established guidelines for surveillance of cancer patients with germline BAP1 mutations or of cancer-free individuals with germline BAP1 mutations.

Objectives:

To prospectively gather information related to the use of dual energy computed tomographic imaging (DECT) together with minimally invasive surgical surveillance for early detection of pleural or peritoneal mesothelioma in participants with BAP1 tumor predisposition syndrome (TPDS)

Eligibility:

* Individuals with a history of any malignancy with known or suspected germline mutation involving BAP1.
* First- or second-degree relatives of patients with documented germline BAP1 mutations, who are also found to carry similar germline mutations.
* Age greater than or equal to 30

Design:

* Participants with suspected hereditary tumor predisposition syndromes will undergo germline evaluation using CLIA-certified next-gen sequencing (NGS).
* First- and second-degree relatives of patients with germline BAP1 mutations who become protocol participants will be offered similar NGS evaluation.
* Participants with germline mutations in BAP1 will undergo periodic dual energy CT (DECT) scans of the chest, abdomen, and pelvis. Plasma cell-free DNA (cfDNA) will be assessed at similar intervals, and minimally invasive surveillance procedures (i.e., video-assisted thoracoscopy and laparoscopy) will be performed periodically to detect early, subclinical malignancies that may be amenable to potentially curative local interventions.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Inclusion Criteria for Genetic Testing

-Eligible participants include:

--Individuals with a history of any malignancy with known or suspected germline mutations involving BAP1

OR

--First- or second-degree relatives of patients (with or without cancer) with documented BAP1 tumor predisposition syndrome (TPDS).

* Age greater than or equal to 30 years.
* All participants must understand and be willing to sign a written informed consent document.

Inclusion Criteria for Surveillance

* Eligible participants include those who completed step 1 genetic testing with study-confirmed BAP1 or other germline TPDS mutation.
* Completed co-enrollment on protocol 06C0014, "Prospective Evaluation of Genetic and Epigenetic Alterations in Patients with Thoracic Malignancies."

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals, and family members of the individual, who fulfill clinical criteria of a history of cancer and detected or suspected germline mutation in BAP1 TPDS.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2038-06-30 (Estimated); Study Completion 2038-06-30 (Estimated)

PRIMARY OUTCOMES:
Prospectively gather information related to the use of dual energy computed tomographic imaging (DECT) together with minimally invasive surveillance for early detection of mesotheliomas in patients with BAP1 TPDS | annual or biennial follow-up, 5 years interim analysis
  Documentation of the counts, incidence, and frequencies of cancers from dual energy computed tomographic imaging and minimally invasive surveillance results will be analyzed for statistical analysis for the early detection of mesotheliomas in patients with BAP1 TPDS.

SECONDARY OUTCOMES:
To characterize the epigenetic features of mesotheliomas associated with germline mutations in BAP1 | at clinical visits, annual or bi-annual follow-up
  Characterization of the epigenetic features of mesotheliomas associated with germline mutations in BAP1.
To investigate the biological mechanisms associated with prolonged survival in participants with mesothelioma that carry germline BAP1 mutations | once during follow-up per participant agreement
  Tumor tissue, blood, saliva, or buccal swab specimen for genetic analyses including WES, FACS, Western blots, and RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0106.html